CLINICAL TRIAL: NCT01447277
Title: The Addition of a Preoperative Sciatic Nerve Block to a Femoral Nerve Block for Ambulatory Arthroscopic ACL Reconstruction
Brief Title: Prospective Femoral Versus Femoral and Sciatic Nerve Block for Anterior Cruciate Ligament (ACL) Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-06776
Record Dates: First submitted 2011-09-30; First posted 2011-10-06 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Anterior Cruciate Ligament Tear
Keywords: ACL reconstruction; Femoral Block; Sciatic Block
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femoral and Sciatic Block (Experimental): Administration of preoperative femoral and sciatic nerve blocks
  Interventions: Procedure: Sciatic Block
- Femoral Block Only (Other): Administration of a femoral nerve block prior to surgery
  Interventions: Procedure: Femoral Block only

INTERVENTIONS:
Procedure: Sciatic Block — Performing a sciatic block in addition to a femoral block preoperatively
  Arms: Femoral and Sciatic Block
Procedure: Femoral Block only — Performing a preoperative sciatic nerve block only
  Arms: Femoral Block Only

SUMMARY:
The investigators propose that a preoperative femoral and sciatic blocks vs a femoral block only, prior to ambulatory anterior cruciate ligament (ACL) reconstruction will lead to a decrease in opiate consumption, pain scores, and post-anesthesia care unit (PACU) length of stay. The investigators are prospectively randomizing patients to either a femoral or a fem/sciatic block and monitor outcomes.

DETAILED DESCRIPTION:
Although femoral nerve blocks improve analgesia after anterior cruciate ligament (ACL) reconstruction, patients often complain of posterior knee pain, which can be treated with a sciatic nerve block. In a prospective randomized study, we compare preoperative femoral nerve block to a combined femoral and sciatic block in patients undergoing ambulatory ACL reconstruction. We hypothesize that the combined femoral/sciatic nerve block patients would have improved analgesia, fewer opioid-related side effects, and shorter PACU length of stay and improved patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* ASA status I-II
* Scheduled for ambulatory Arthroscopic ACL Surgery

Exclusion Criteria:

* Allergy to Local anesthetics or opiates used in the study
* Contraindications for regional anesthesia
* coagulopathy, anticoagulation, Thrombocytopenia
* infection at site of injection
* Chronic pain and high preoperative opiate requirements
* High risk for PONV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Pain Scores | PACU and POD1, 2 and 3.

SECONDARY OUTCOMES:
Length of stay | Duration of stay in the recovery room
Opiate consumption | During surgery, recovery room and for 3 days after discharge
PONV | During the recovery room stay and after discharge from surgery center for up to 3 days.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Orthopedic Institute, San Francisco, California, United States